CLINICAL TRIAL: NCT05134636
Title: Text-based Intervention to Minimize the Time Burden of Routine Cancer Care
Acronym: TIME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UPCC 16921
Record Dates: First submitted 2021-11-15; First posted 2021-11-26 (Actual); Results first posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Cancer; Solid Tumor; Patient Empowerment; Telemedicine
MeSH Terms: conditions — Neoplasms; Patient Participation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Experimental): For patients in the intervention arm, symptoms and laboratory results will be assessed using the text-based e-triage 96 hours prior to their intended infusion date. The e-triage will consist of a standardized questionnaire and algorithm to evaluate symptoms and laboratory values. Patients with acceptable labs and minimal or no symptoms can opt to proceed directly to their immunotherapy infusion without an in-person office assessment.
  Interventions: Other: Text triage
- Usual Care (No Intervention): Patients in the usual care arm will receive standard of care symptom monitoring including an in-person office assessment prior to their scheduled immunotherapy infusion.

INTERVENTIONS:
Other: Text triage — The e-triage will consist of 16 questions, modified from the validated NCI Pro-CTCAETM, which will be sent to patients via WaytoHealth©'s two-way texting system 96 hours prior to their scheduled immunotherapy infusion. Questions will pertain to common or emergent immune related adverse events as defined by the NCCN guidelines and two senior disease experts. Patients will be prompted via text to measure the presence and severity of symptoms over the week prior. A final question will be included to capture any additional symptoms patients wish to disclose.
  Arms: Treatment Arm

SUMMARY:
The primary objective is to test whether a text-based e-triage can safely minimize the time associated with routine cancer care by identifying patients who can proceed directly to their immunotherapy infusion without a preceding in-person office assessment.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Initiating singe agent PDL-1/PD-1 targeted immune checkpoint blockade for any solid malignancy at Penn's Abramson Cancer Center
* Access to a mobile phone with texting capabilities
* ECOG performance status less than or equal to 2

Exclusion Criteria:

* Non-English speaking
* Unable to perform informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin Bange, MD, Principal Investigator — Fellow; Ronac Mamtani, MD, MSCE, Principal Investigator — Faculty
Locations (1):
- Perelman Center for Advanced Care, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in publication, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: IPD will be shared with researchers who provide a methodologically sound proposal, for the purpose of achieving aims in the approved proposal. Proposals should be directed to bangee@mskcc.org and ronac.mamtani@pennmedicine.upenn.edu. To gain access, data requestors will need to sign a data access agreement. Data will be available upon request.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Run-in period during which patients were sent a preliminary text message asking them to confirm study participation. 11 patients did not respond to this enrollment text.
Period: Overall Study
Arm/Group | Treatment Arm | Usual Care
Started | 19 | 21
Completed | 16 | 15
Not Completed | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Arm | Usual Care | Total
Number analyzed (Participants) | 19 | 21 | 40
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 67 [62 to 74] | 69 [59 to 71] | 67 [59.5 to 71.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 16 | 16 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 14 | 20 | 34
  Unknown or Not Reported | 4 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 14 | 19 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Distance in Miles from Cancer Center [Number; unit: participants]
  0-19.3 miles | 6 | 3 | 9
  19.31-33.13 miles | 4 | 5 | 9
  33.14-49.38 miles | 4 | 5 | 9
  49.39-150 miles | 4 | 4 | 8
  Missing | 1 | 4 | 5
Marital Status [Count of Participants; unit: Participants]
  Single | 1 | 2 | 3
  Married | 16 | 15 | 31
  Divorced | 1 | 2 | 3
  Widowed | 0 | 2 | 2
  Missing | 1 | 0 | 1
Highest Education [Count of Participants; unit: Participants]
  High school diploma/GED | 3 | 6 | 9
  Technical or trade school | 3 | 1 | 4
  Some college | 3 | 2 | 5
  Associate degree | 2 | 1 | 3
  Bachelor's degree | 3 | 5 | 8
  Some graduate school | 1 | 1 | 2
  Master's degree | 3 | 5 | 8
  Unknown | 1 | 0 | 1
Income [Count of Participants; unit: Participants]
  $0-20,000 | 2 | 2 | 4
  $20,001-40,000 | 2 | 2 | 4
  $40,001-60,000 | 0 | 3 | 3
  $60,001-80,000 | 1 | 4 | 5
  $80,001-100,000 | 0 | 2 | 2
  $100,001+ | 11 | 5 | 16
  Missing | 3 | 3 | 6
Tumor Stage [Count of Participants; unit: Participants] — Cancer staging describes the severity of an individual's cancer based on the magnitude of the original (primary) tumor as well as on the extent cancer has spread in the body, and is determined by the patient's primary oncologist, with 1 being least severe.
  Participants
    1 | 0 | 1 | 1
    2 | 1 | 0 | 1
    3 | 7 | 4 | 11
    4 | 9 | 16 | 25
    Missing | 2 | 0 | 2
Tumor Type [Count of Participants; unit: Participants]
  Genitourinary | 10 | 14 | 24
  Thoracic | 4 | 5 | 9
  Skin | 3 | 0 | 3
  Head and Neck | 2 | 0 | 2
  Gastrointestinal | 0 | 1 | 1
  Other | 0 | 1 | 1
ICI Type [Count of Participants; unit: Participants]
  Pembrolizumab | 13 | 17 | 30
  Nivolumab | 2 | 2 | 4
  Avelumab | 1 | 1 | 2
  Atezolizumab | 1 | 1 | 2
  Cemiplimab | 1 | 0 | 1
  Durvalumab | 1 | 0 | 1
Lines of Prior Therapy [Count of Participants; unit: Participants]
  0 | 12 | 9 | 21
  1 | 4 | 10 | 14
  2 | 0 | 2 | 2
  3+ | 3 | 0 | 3
Patient-reported ECOG PS [Count of Participants; unit: Participants] — The ECOG Performance Status Scale describes a patient's self-reported level of functioning in terms of their ability to care for themselves, daily activity, and physical ability (walking, working, etc.).
  0 Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities
  3. Capable of only limited selfcare
  4. Completely disabled
  5. Dead
  Participants
    0-1 | 12 | 14 | 26
    2+ | 4 | 2 | 6
    Missing | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Healthcare Time
Description: Time spent commuting to, waiting for, and receiving healthcare over a 3 month follow up period.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Treatment Arm | Usual Care
Number analyzed (Participants) | 19 | 21
minutes | 265.97 (77.6) | 339.54 (108.29)

2. Secondary Outcome: Total Wait Time
Description: Time spent waiting for healthcare over a 3 month follow up period.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Treatment Arm | Usual Care
Number analyzed (Participants) | 19 | 21
minutes | 124.79 (44.35) | 154.71 (72.34)

3. Secondary Outcome: Total Number of Hospitalization/Emergency Department Encounters
Description: Total number of hospitalizations and emergency department encounters over a 3 month follow up.
Time Frame: 3 months
Measure: Number; unit: admissions
Arm/Group | Treatment Arm | Usual Care
Number analyzed (Participants) | 19 | 21
admissions | 3 | 2

4. Secondary Outcome: Patient Satisfaction as Assessed by the Patient Satisfaction Questionnaire Short Form (PSQ-18)
Description: The Patient Satisfaction Questionnaire Short Form (PSQ-18) is a self-reported measure capturing satisfaction with medical care across 7 dimensions, all subscales (no total).
  * General Satisfaction (3&17) - higher scores represent greater satisfaction
  * Technical Quality (2, 4, 6, 14) -higher scores represent better technical quality
  * Interpersonal Manner (10&11) - higher scores represent better interpersonal manner
  * Communication (1&13) - higher scores represent better communication
  * Financial Aspects (5&7) - higher scores represent better financial aspects
  * Time Spent with Doctor (12&15) - higher scores represent better time spent w/ dr
  * Accessibility and Convenience (8, 9, 16, 18) - higher scores represent more accessibility Reverse scoring takes place for items 1, 2, 3, 5, 6, 8, 11, 15, and 18 such that a response of 1 has a score value of 5, and so on.
  After noting score values for each individual response, items are then averaged for each subscale to gain a subscale score.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale of 5
Arm/Group | Treatment Arm | Usual Care
Number analyzed (Participants) | 19 | 21
units on a scale of 5
  General Satisfaction (0-5) | 4.34 (.59) | 4.5 (0.77)
  Technical Quality (0-5) | 4.42 (0.77) | 4.48 (0.58)
  Interpersonal Manner (0-5) | 4.19 (0.77) | 4.64 (0.41)
  Communication (0-5) | 4.25 (0.86) | 4.61 (0.45)
  Financial Aspects (0-5) | 3.88 (0.87) | 3.82 (0.77)
  Time Spent with Doctor (0-5) | 4.38 (0.59) | 4.32 (0.64)
  Accessibility and Convenience (0-5) | 3.72 (0.58) | 3.93 (0.58)

5. Secondary Outcome: Health Related Quality of Life as Assessed by the Functional Assessment of Cancer Therapy-General (FACT-G)
Description: The Functional Assessment of Cancer Therapy-General (FACT-G) is a 27-item questionnaire comprised of four subscales to measure health-related quality of life:
  * physical well-being (PWB; 7-items, score range 0-28), higher score = better PWB
  * social/family well-being (SWB; 7-items, score range 0-28), higher score = worse SWB
  * emotional well-being (EWB; 6-items, score range 0-24), higher score = better EWB except item 2 where higher score = worse EWB
  * functional well-being (FWB; 7-items, score range 0-28), higher score = worse FWB All questions in the FACT-G use a 5-point rating scale (0=Not at all; 1=A little bit; 2=Somewhat; 3=Quite a bit; 4=Very much). Within a subscale, response are reversed for those where higher score = worse well-being, and then averaged for the scale score.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Arm | Usual Care
Number analyzed (Participants) | 19 | 21
units on a scale
  Physical well-being (0-28) | 23.21 (5.31) | 23.4 (4.27)
  Social/family well-being (0-28) | 22.48 (5.04) | 25.71 (5.39)
  Emotional well-being (0-24) | 17.66 (5.45) | 20.6 (3)
  Functional well-being (0-28) | 17.19 (9) | 21 (4.24)

ADVERSE EVENTS:
Time Frame: 3 months
Description: Minimal risk study - adverse events as defined did not result from our intervention
Arm/Group | Treatment Arm | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/21
Other Adverse Events (participants affected / at risk) | 0/19 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-03-01): https://cdn.clinicaltrials.gov/large-docs/36/NCT05134636/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-01): https://cdn.clinicaltrials.gov/large-docs/36/NCT05134636/SAP_001.pdf